CLINICAL TRIAL: NCT07355673
Title: A Double Blind Randomized Clinical Trial Comparing the Risk of Gingival Irritation of Two Different Isolation Techniques Performed During In-Office Bleaching
Brief Title: The Influence of Isolation Techniques in Gingival Irritation During an In-office Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Patricia Pereira-Lores, Principal Investigator, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025/02
Record Dates: First submitted 2025-12-10; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Gingival Irritation
Keywords: Gingival irritation; Vital Bleaching; In-Office bleaching; Isolation

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Clinical Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Relative Isolation (Active Comparator): The relative isolation technique consists in inserting a lip retractor (OptraGate, Ivoclar Vivadent) and applying a gingival barrier resin (OpalDam, Ultradent Products) along the gingival margin, extending approximately 2-3 mm onto the enamel.
  Interventions: Device: Relative Isolation
- Absolute isolation (Experimental): The total rubber dam isolation was carried out placing the dam (Flexidam non latex; Roeko) from premolar to premolar in both arches and stabilizing it with clamps (B4; Hygenic). Dental silk ligatures were used to achieve proper cervical retraction.
  Interventions: Device: Absolute Isolation

INTERVENTIONS:
Device: Relative Isolation — General Examination with bite-wings, dental prophylaxis, alginate impressions of both arches, creation of individualized bleaching trays and position finder trays. . Relative isolation of the gingival tissues. Two applications of the bleaching agent of 20 minutes
  Arms: Relative Isolation
Device: Absolute Isolation — General Examination with bite-wings, dental prophylaxis, alginate impressions of both arches, creation of individualized bleaching trays and position finder trays. . Absolute isolation of the gingival tissues. Two applications of the bleaching agent of 20 minutes
  Arms: Absolute isolation

SUMMARY:
The objective of this study was to evaluate if two different isolation techniques used during in-office bleaching influence the risk of gingival irritation. The secondary objectives were to investigate whether the isolation technique affects bleaching efficacy, the occurrence of tooth sensitivity, and the intensity of tooth sensitivity (TS).

DETAILED DESCRIPTION:
1. Visit 1: Study information and delivery of informed consent. Recording of patient's medical history, general examination, and prophylaxis. Alginate impressions will be taken of the upper and lower arches for all the patients who meet the inclusion criteria. The impressions will be poured into plaster, and a positioning guide-finder tray will be fabricated for each patient for color measurement.
2. Visit 2: Initial color measurement with a spectrophotometer and the positioning guide. Two clinicians performed the assigned isolation technique (relative or absolute). Then after a correct isolation the clinicians apply over the buccal surface from premolar to premolar of both arches the bleaching agent (Opalescence Boost 40%, Ultradent Products, South Jordan, USA).Two application of 20 minutes each. Objective examination of gingival tissues was performed visually, documented with photographs, and verified using a periodontal probe. The sensitivity was recorded and patient were given a sensitivity test to record at home. c) Visit 3: One week after the first bleaching session. Color measurement with a spectrophotometer and the positioning guide. In this visit the second bleaching session was done with the same steps as visit 2. d) Visit 4: 15 days after the second bleaching session. Final data collection (color + patients sensitivity test)

ELIGIBILITY:
Inclusion Criteria:

* No oral os systemic pathology
* Periodontally Healthy
* No cavities
* Tooth shade of the canines A2 or darker

Exclusion Criteria:

* Adhesive restorations or protheses in the anterior region
* Enamel or dentin alterations
* Smoking habits
* Pregnant women
* Undergone prior bleaching treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Gingival Evaluation Recording | -15 minutes after the first bleaching session - 15 minutes after the second bleaching session
  Objective examination of gingival tissues was performed visually, documented with photographs, and verified using a periodontal probe. Patients were classified according to the Löe and Silness' gingival index as follows: G0 =normal gingiva; G1=mild inflammation (slight color change, slight edema, no bleeding on probing); G2=moderate inflammation (redness, edema, glazing, bleeding on probing); and G3=severe inflammation (marked redness and edema, ulceration, spontaneous bleeding).

SECONDARY OUTCOMES:
Questionary of dental sensitivity | Perioperative , 1 hour postoperative, 24 hours postoperative, 48 hours postoperative.
  General tooth sensitivity was assessed using a 5-point Numeric Rating Scale (NRS), where 0 = no sensitivity; 1 = mild discomfort; 2 = moderate discomfort that does not interfere with daily activities; 3 = considerable discomfort leading to avoidance of certain foods and beverages; and 4 = severe sensitivity requiring interruption of the bleaching treatment. Participants selected the numeric value that best represented their perceived level of tooth sensitivity.
  Pain intensity was recorded at the following time points:
  * Perioperative
  * 1 hour postoperatively
  * 24 hours postoperatively
  * 48 hours postoperatively
Shade evaluation of each patient | Baseline, Before the first bleaching session, Revision (1 week after the 2 bleaching session)
  Tooth color will be measured using a dental spectrophotometer, recording the following parameters: L (lightness, representing the shade from black to white on a scale of 0 to 100), a (color variation along the red-green axis, with positive values toward red/purple and negative values toward green/blue), b (color variation along the yellow-blue axis, with positive values toward yellow and negative values toward blue/purple), C (chroma, describing the intensity or saturation of a color, expressed on a scale from 0 to 40, where 0 indicates no saturation and 40 the maximum saturation), and hº (hue, representing the dominant wavelength of a color on a continuous circular scale from 0° to 360°).
  Color changes between visits will be calculated using the CIELab, CIEDE2000, and White Index for Dentistry (WID) formulas.
  Color measurements will be recorded at the following time points:
  Baseline (Bleaching Day 1) One week after baseline (Before Bleaching Day 2) Follow-up (One week after)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine and Dentistry, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No